CLINICAL TRIAL: NCT00151437
Title: A Multi-Center, Open-Label Study For The Compassionate Use Of Pegvisomant In Acromegalic Patients Refractory To Conventional Therapy and For Patients Who Received The Product During The Clinical Development Program.
Brief Title: Canadian Pegvisomant Compassionate Study In Acromegalic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6291017
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Health Records, Personal; Demography; Glucose Tolerance Test

INTERVENTIONS:
Drug: Pegvisomant treatment
Procedure: Medical History, demographics
Procedure: Sign and symptoms: questionnaire
Procedure: Blood tests: IGF-1, AST/ALT/ALP/TBIL, GTT
Procedure: MRI

SUMMARY:
The purposes of this study are: 1) to provide SOMAVERT for compassionate use to patients with acromegaly or who have completed clinical trials and were responsive, and 2) to evaluate the safety and tolerability of SOMAVERT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have participated and completed the previous Pegvisomant studies or have shown to be unresponsive to other conventional therapies

Exclusion Criteria:

* ALT/AST>3 times the ULN or have hepatic disease
* have severe visual field loss, cranial nerve palsies or intracranial HTN that requires surgery to decompress the tumor
* unwilling to self-administer the medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-11; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Patient's IGF-1 levels normalize signs and symptoms of acromegaly normalize

SECONDARY OUTCOMES:
Pegvisomant demonstrates continued safety and efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Canada (4):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec

REFERENCES:
- [Derived] Ezzat S, Gaspo R, Serri O, Ur E, Chik CL. A Canadian multi-centre, open-label long-term study of Pegvisomant treatment in refractory acromegaly. Clin Invest Med. 2009 Dec 1;32(6):E265. doi: 10.25011/cim.v32i6.10662. PMID 20003832
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6291017&StudyName=Canadian%20Pegvisomant%20Compassionate%20Study%20In%20Acromegalic%20Patients%20